CLINICAL TRIAL: NCT05816733
Title: Dapagliflozin Evaluation on Atrial Fibrillation Patients Followed Cox Maze IV Procedure: Prospective Randomized Trial (DETAIL-CMIV)
Brief Title: Dapagliflozin Evaluation on Atrial Fibrillation Patients Followed Cox Maze IV Procedure
Acronym: DETAIL-CMIV
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kun Hua (Other)
Responsible Party: Sponsor-Investigator, Kun Hua, Clinical Professor, Beijing Anzhen Hospital
Organization: Beijing Anzhen Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KS2023017
Record Dates: First submitted 2023-04-02; First posted 2023-04-18 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Atrial Fibrillation Recurrence; Cox Maze IV; Atrial Fibrillation; Patients With or Without Heart Failure and Diabetes
MeSH Terms: conditions — Atrial Fibrillation; Diabetes Mellitus | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dapagliflozin group (Experimental): Patients who will be randomized to receive dapagliflozin following the Cox-Maze IV Procedure.
  Interventions: Drug: Dapagliflozin
- Placebo group (Placebo Comparator): Patients who will be randomized to receive placebo following the Cox-Maze IV Procedure.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin — Patients randomized in this arm will receive dapagliflozin at a target dose of 10mg once daily and routine treatment.
  Arms: Dapagliflozin group
Drug: Placebo — Patients randomized in this arm will receive placebo at a target dose of 10mg once daily and routine treatment.
  Arms: Placebo group

SUMMARY:
Atrial fibrillation (AF) is the most common arrhythmia, which leads to reduced cardiac output and promotes the occurrence of heart failure, and abnormal hemodynamic changes in the left atrium induce thrombosis, which seriously reduces the quality of life, and even leads to death. For patients who need cardiac surgery combined with the Cox-Maze IV (CMIV) surgical ablation, oral amiodarone postoperatively for three consecutive months was recommended as the preferred treatment option. However, the study found there were still 15%-35% of patients at risk of AF recurrence. Dapagliflozin, a sodium-glucose cotransporter 2 inhibitor, has been widely used for the treatment of type 2 diabetes mellitus and heart failure. Nonetheless, it remains unknown whether dapagliflozin can improve the recurrence of AF and reduces adverse cardiovascular events for patients who need CMIV ablation, and whether it can be routinely used for AF patients without diabetes or heart failure. Therefore, this study aims to explore the effect of postoperative oral dapagliflozin on the recurrence of AF after CMIV.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Patients with persistent or long-term persistent atrial fibrillation who need isolated surgical Cox-Maze IV procedure
* Patients who need cardiac surgery combined with Cox-Maze IV procedure
* Patients who have the ability and willingness to abide by all the subsequent reviews and requirements
* Sign the informed consent

Exclusion Criteria:

* Dapagliflozin allergy
* Hyperthyroidism
* Patients with acute myocardial infarction, cerebral apoplexy, and other vascular diseases during the past 6 months
* Patients who received heart surgery within the last 3 months
* eGFR<45ml/min
* History of oral SGLT2i
* Estimated survival period < 12 months
* Pregnant and lactating women
* Left atrial diameter > 65 mm
* Refusing to sign the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 348 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-06-07 (Estimated); Study Completion 2024-08-07 (Estimated)

PRIMARY OUTCOMES:
Rate of atrial fibrillation recurrence | half of one year post operative

SECONDARY OUTCOMES:
Rate of atrial fibrillation recurrence | one year post operative
Cardiovascular complex adverse events | one year post operative
  cardiogenic death, new onset heart failure, malignant arrhythmias, stroke

CONTACTS AND LOCATIONS:
Overall Officials: Kun Hua, Study Director — Beijing Anzhen Hospital
Locations (1):
- Cardiac Surgery Center No. 7, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided